CLINICAL TRIAL: NCT02120950
Title: A Randomized, Double-masked, Sham-controlled Phase 3b/4 Study of the Efficacy, Safety, and Tolerability of Intravitreal Aflibercept Monotherapy Compared to Aflibercept With Adjunctive Photodynamic Therapy as Indicated in Subjects With Polypoidal Choroidal Vasculopathy
Brief Title: Aflibercept in Polypoidal Choroidal Vasculopathy
Acronym: PLANET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16995; 2013-004464-54 (EudraCT Number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-23 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Neovascular Macular Degeneration
Keywords: PCV
MeSH Terms: interventions — aflibercept; Verteporfin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept + Sham PDT (Experimental): Participants received 2 milligram (mg) Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period). At Week 12, subjects were randomized to receive Aflibercept injection plus sham photodynamic therapy (only in subjects qualifying for rescue therapy)
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Aflibercept + Active PDT (Experimental): Participants received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period). At Week 12, subjects were randomized to receive Aflibercept injection plus active photodynamic therapy (only in subjects qualifying for rescue therapy)
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321); Other: Visudyne

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Eylea is administered as an intravitreal injection
Other: Visudyne — Photodynamic therapy is a combined therapy of drug (Visudyne) applied to reinforce the action of a device (laser)
  Arms: Aflibercept + Active PDT

SUMMARY:
To collect data reflecting the efficacy and safety of aflibercept with and without photodynamic therapy in subjects diagnosed with the polypoidal choroidal vasculopathy subtype of wet age-related macular degeneration

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men and women ≥50 years of age
* Diagnosis of symptomatic macular Polypoidal Choroidal Vasculopathy (PCV) in the study eye established by Indocyanine Green Angiography(ICGA) at the study center
* Greatest linear dimension of the lesion of < 5400 mm (approximately, 9 Macular Photocoagulation Study disk areas), assessed by ICGA.
* An Early treatment diabetic retinopathy study (ETDRS) BCVA of 73 to 24 letters in the study eye.

Exclusion Criteria:

* Prior use of intravitreal or sub-tenon corticosteroids in the study eye within 3 months prior to study entry
* Any prior use of intraocular anti Vascular Endothelial Growth Factor (anti-VEGF)agents in the study eye, or systemic use of anti VEGF products within 3 months prior to study entry
* Prior macular laser treatment in the study eye including Photodynamic Therapy (PDT)
* History of allergy to fluorescein used in fluorescein angiography, iodine and/or indocyanine green.
* History of allergy to aflibercept, verteporfin, or their excipients.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (49):
- Australia (5):
  - Liverpool, New South Wales
  - Strathfield, New South Wales
  - Westmead, New South Wales
  - East Melbourne, Victoria
  - Parramatta
- München, Germany
- Hong Kong (2):
  - Hong Kong
  - Kowloon
- Hungary (2):
  - Budapest
  - Debrecen
- Japan (33):
  - Nagoya, Aichi-ken
  - Urayasu, Chiba
  - Ōgaki, Gifu
  - Maebashi, Gunma
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - Kobe, Hyōgo
  - Kita, Kagawa-ken
  - Tsu, Mie-ken
  - Kashihara, Nara
  - Hirakata, Osaka
  - Suita, Osaka
  - Ōtsu, Shiga
  - Hamamatsu, Shizuoka
  - Shimotsuke, Tochigi
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Meguro-ku, Tokyo
  - Mitaka, Tokyo
  - Shinjuku-ku, Tokyo
  - Akita
  - Aomori
  - Chiba
  - Fukuoka
  - Fukushima
  - Kumamoto
  - Kyoto
  - Nagasaki
  - Okayama
  - Osaka
  - Tokushima
  - Wakayama
- Singapore, Singapore
- South Korea (2):
  - Seongnam-si, Gyeonggido
  - Seoul
- Taiwan (3):
  - Changhua, Changhua
  - Kaohsiung City
  - Taipei

REFERENCES:
- [Derived] Lee WK, Iida T, Ogura Y, Chen SJ, Wong TY, Mitchell P, Cheung GCM, Zhang Z, Leal S, Ishibashi T; PLANET Investigators. Efficacy and Safety of Intravitreal Aflibercept for Polypoidal Choroidal Vasculopathy in the PLANET Study: A Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jul 1;136(7):786-793. doi: 10.1001/jamaophthalmol.2018.1804. PMID 29801063
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=16995&attachmentIdentifier=6557dbc1-0000-454b-9bbc-69a823522784&fileName=16995_Study_Synopsis_CTP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 8 countries worldwide starting from 29 May 2014 (first subject first visit). Primary completion reached on 12 Aug 2016.
Pre-assignment Details: Overall, 428 subjects were screened, of them 95 were failed in screening. Remaining 333 subjects received at least one treatment. Of them, 15 subjects discontinued study participation before week 12 and were not randomized. Remaining 318 were randomized.
Groups:
- Aflibercept + Sham Photodynamic Therapy (PDT): Participants received 2 milligram (mg) Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period). At Week 12, subjects were randomized to receive Aflibercept injection plus sham photodynamic therapy (only in subjects qualifying for rescue therapy).
- Aflibercept + Active PDT: Participants received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period). At Week 12, subjects were randomized to receive Aflibercept injection plus active photodynamic therapy (only in subjects qualifying for rescue therapy) until Week 52. Between Week 52 and Week 96, the treatment interval could have been extended (typically in increments of 1 or 2 weeks) at the discretion of the investigator when the visual and anatomic outcomes allowed
- Aflibercept (Non-randomized): Participants received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period), but discontinued study participation before randomization
Period: Overall Study
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT | Aflibercept (Non-randomized)
Started | 157 | 161 | 15
Completed | 137 (Completed Treatment (Week 96)) | 147 (Completed Treatment (Week 96)) | 0
Not Completed | 20 | 14 | 15
Not completed — Adverse Event | 5 | 4 | 3
Not completed — Death | 3 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 2
Not completed — Protocol Violation | 1 | 1 | 7
Not completed — Other reasons | 5 | 4 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics is reported in Full analysis set which included all randomized subjects (N=318).
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT | Total
Number analyzed (Participants) | 157 | 161 | 318
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.8 (8.4) | 70.4 (8.0) | 70.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 49 | 96
  Male | 110 | 112 | 222
Baseline BCVA score [Mean (Standard Deviation); unit: Letters] — Visual function of the study eye and fellow eye was assessed at each study visit according to the standard procedure developed for the ETDRS adapted for AREDS, using 70 letter charts at a starting distance of 4 meters. Participants were challenged with reading letters on lines of an eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until they reached a row where a minimum of three letters on a line could be read, and were scored by how many letters could be correctly identified.
  Letters | 57.7 (11.3) | 59.0 (11.5) | 58.4 (11.4)
Central Subfield Thickness [Mean (Standard Deviation); unit: Micrometer] | 347.8 (118.9) | 346.1 (117.5) | 346.9 (118.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment of Diabetic Retinopathy Study (ETDRS) Letter Scores From Baseline to Week 52 - Last Observation Carried Forward (LOCF)
Description: Visual function of the study eye and fellow eye was assessed at each study visit according to the standard procedure developed for the ETDRS adapted for Age Related Eye Disease Study (AREDS), using 70 letter charts at a starting distance of 4 meters. Participants were challenged with reading letters on lines of an eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until they reached a row where a minimum of three letters on a line could be read, and were scored by how many letters could be correctly identified.
Time Frame: From Baseline to Week 52
Population: Full Analysis Set (FAS) included all randomized subjects
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Letters correctly read | 10.7 (11.3) | 10.8 (10.7)
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Test type: Superiority or Other; p = 0.5480, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.9 to 1.6]

2. Secondary Outcome: Percentage of Subjects Who Avoided at Least 15 Letters Loss in ETDRS at Week 52
Description: as for outcome 1
Time Frame: At Week 52
Population: FAS
Measure: Number; unit: Percentage of subjects
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Percentage of subjects | 97.5 | 96.9
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Test type: Superiority or Other; p = 0.7402, Cochran-Mantel-Haenszel; treatment difference in % = 0.6, 95% CI 2-sided [-3.1 to 4.3]

3. Other Pre Specified Outcome: Percentage of Subjects Who Never Need Rescue Therapy in the First Year
Description: Evaluations for qualification for rescue were conducted at each visit from Week 12 to Week 52. Intensified aflibercept treatment plus active or sham PDT treatments were given at any of these visits if treatment criteria were met. Qualification for rescue was based upon insufficient gain of BCVA, leakage, and presence of active polyps.
Time Frame: Baseline to Week 52
Population: FAS
Measure: Number; unit: Percentage of subjects
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Percentage of subjects | 87.9 | 85.7

4. Other Pre Specified Outcome: Number of PDT Treatments in the Study Eye Before Week 52
Time Frame: Baseline to Week 52
Population: FAS
Measure: Mean (Standard Deviation); unit: PDT administrations
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
PDT administrations | 0.2 (0.7) | 0.2 (0.4)
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Test type: Superiority or Other; p = 0.0682, ANCOVA; LS mean difference = 0.1, 95% CI 2-sided [0.0 to 0.2] — Point estimate, 95% CI and p-value are based on treatment difference (AFL-sham - AFL-PDT) of the LS mean changes using an ANOVA model with treatment group and ethnicity and qualification for rescue therapy at Week 12 as fixed effects

5. Other Pre Specified Outcome: Number of Aflibercept Treatments in the Study Eye (After Randomization) Before Week 52
Time Frame: Baseline to Week 52
Population: FAS with evaluable subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: Aflibercept injections
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 154 | 160
Aflibercept injections | 5.2 (1.1) | 5.1 (0.8)
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Test type: Superiority or Other; p = 0.1640, ANCOVA; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.3] — [estimate comment as in outcome 4, analysis 1]

6. Other Pre Specified Outcome: Time to First Administration of PDT in the Study Eye Before Week 52
Time Frame: Baseline to Week 52
Population: FAS
Measure: Mean (Full Range); unit: Days
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Days | 131.2 [80 to 278] | 128.2 [80 to 315]

7. Other Pre Specified Outcome: Change of Visual Acuity (Letters) From Baseline Over Time (Week) in the Study Eye
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: FAS
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Letters | 10.7 (11.3) | 10.8 (10.7)

8. Other Pre Specified Outcome: Percentage of Subjects Who Gained ≥5, 10, or 15 Letters at Week 52
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: FAS
Measure: Number; unit: Percentage of subjects
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Percentage of subjects
  Gained ≥ 5 | 73.9 | 78.9
  Gained ≥ 10 | 55.4 | 57.1
  Gained ≥ 15 | 33.1 | 36.6
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Category of Gained ≥ 5; Test type: Superiority or Other; p = 0.2348, Cochran-Mantel-Haenszel; The p-value is calculated from the 2-sided Cochran-Mantel-Haenszel test adjusted by ethnicity and qualification for rescue therapy at Week 12; treatment difference in % = -5.6, 95% CI 2-sided [-14.9 to 3.7] — CI is based on the treatment difference in % (AFL-sham - AFL-PDT) using the Mantel-Haenszel weighting scheme adjusted by ethnicity and qualification for rescue therapy at Week 12
Statistical Analysis 2: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Category of Gained ≥ 10; Test type: Superiority or Other; p = 0.6877, Cochran-Mantel-Haenszel; [statistical method as in outcome 8, analysis 1]; treatment difference in % = -2.2, 95% CI 2-sided [-13.1 to 8.6] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Category of Gained ≥ 15; Test type: Superiority or Other; p = 0.4556, Cochran-Mantel-Haenszel; [statistical method as in outcome 8, analysis 1]; treatment difference in % = -4.0, 95% CI 2-sided [-14.5 to 6.5] — [estimate comment as in outcome 8, analysis 1]

9. Other Pre Specified Outcome: Percentage of Subjects Who Lost ≥5, 10, or 15 Letters at Week 52
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: FAS
Measure: Number; unit: Percentage of subjects
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Percentage of subjects
  Lost ≥ 5 | 7.0 | 5.6
  Lost ≥ 10 | 3.8 | 3.1
  Lost ≥ 15 | 2.5 | 3.1
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Category of Lost ≥ 5; Test type: Superiority or Other; p = 0.5372, Cochran-Mantel-Haenszel; [statistical method as in outcome 8, analysis 1]; treatment difference in % = 1.7, 95% CI 2-sided [-3.7 to 7.2] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Category of Lost ≥ 10; Test type: Superiority or Other; p = 0.7569, Cochran-Mantel-Haenszel; [statistical method as in outcome 8, analysis 1]; treatment difference in % = 0.6, 95% CI 2-sided [-3.4 to 4.7] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Category of Lost ≥ 15; Test type: Superiority or Other; p = 0.7402, Cochran-Mantel-Haenszel; [statistical method as in outcome 8, analysis 1]; treatment difference in % = -0.6, 95% CI 2-sided [-4.3 to 3.1] — [estimate comment as in outcome 8, analysis 1]

10. Other Pre Specified Outcome: Percentage of Subjects With Complete Polyp Regression at Week 52
Description: Complete polyp regression was defined as absent or indeterminate visual polyps on Indocyanine green angiography (ICGA) in the study eye.
Time Frame: Baseline to Week 52
Population: FAS with evaluable subjects for this outcome measure.
Measure: Number; unit: Percetage of subjects
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 126 | 134
Percetage of subjects | 38.9 | 44.8
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Test type: Superiority or Other; p = 0.3244, Cochran-Mantel-Haenszel; [statistical method as in outcome 8, analysis 1]; treatment difference in % = -6.0, 95% CI 2-sided [-17.8 to 5.9] — [estimate comment as in outcome 8, analysis 1]

11. Other Pre Specified Outcome: Change of Leakage Area in Fluorescein Angiography (FA) in the Study Eye at Week 52
Description: Leakage is the release of fluorescein dye from diseased retinal vessels. Leakage area is defined as the area showing presence of fluorescein dye in the late stages of fluorescein angiography.
Time Frame: Baseline to Week 52
Population: FAS with evaluable subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: Square millimeter
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 140 | 149
Square millimeter | -1.3 (3.6) | -1.2 (3.7)
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; The analysis population included only subjects with leakage in FA at baseline and Week 52. Baseline values were not carried forward; Test type: Superiority or Other; p = 0.7109, ANCOVA; LS mean difference = -0.1, 95% CI 2-sided [-0.9 to 0.6] — Point estimate, 95% CI and p-value are based on difference (AFL-sham - AFL-PDT) of LS mean changes using an ANCOVA model with treatment group and ethnicity and qualification for rescue therapy at Week 12 as fixed effects, baseline value as covariate

12. Other Pre Specified Outcome: Change of Central Subfield Thickness (CST) on Optical Coherence Tomography (OCT) From Baseline to Week 52
Description: Retinal and lesion characteristics, such as central retinal thickness (CRT), were evaluated by OCT in both eyes at every study visit. CRT was measured using optical coherence tomography to determine the average thickness of the retina in a circle with 1 millimeter of diameter centered on the fovea. This value is reported by some OCT devices as central subfield thickness (CST).
Time Frame: Baseline to Week 52
Population: FAS with evaluable subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 136 | 150
Millimeter | -137.7 (116.0) | -143.5 (110.5)
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; The analysis population included only subjects with values for CST at baseline and Week 52. Baseline values were not carried forward; Test type: Superiority or Other; p = 0.8355, ANCOVA; LS mean difference = 1.1, 95% CI 2-sided [-9.2 to 11.3] — [estimate comment as in outcome 11, analysis 1]

13. Other Pre Specified Outcome: Change in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Total Score From Baseline to Week 52
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
Time Frame: Baseline to Week 52
Population: FAS with evaluable subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 143 | 153
Scores on a scale | 4.7 (10.3) | 7.3 (12.5)
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; The analysis population included only subjects with values for NEI VFQ-25 score at baseline and Week 52; Test type: Superiority or Other; p = 0.5069, ANCOVA; LS mean difference = -0.7, 95% CI 2-sided [-2.9 to 1.4] — [estimate comment as in outcome 11, analysis 1]

14. Other Pre Specified Outcome: Percentage of Subjects for Whom Rescue Therapy is Indicated Over the Course Till Week 52
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: FAS with evaluable subjects for this outcome measure.
Measure: Number; unit: Percentage of subjects
Arm/Group | Aflibercept + Sham Photodynamic Therapy (PDT) | Aflibercept + Active PDT
Number analyzed (Participants) | 157 | 161
Percentage of subjects | 12.1 | 14.3
Statistical Analysis 1: Comparison: Aflibercept + Sham Photodynamic Therapy (PDT) vs Aflibercept + Active PDT; Test type: Superiority or Other; p = 0.8423, Cochran-Mantel-Haenszel — The p-value is calculated from the 2-sided Cochran-Mantel-Haenszel test adjusted by ethnicity and qualification for rescue therapy at Week 12; Difference % = -0.6, 95% CI 2-sided [-6.3 to 5.1] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after the last treatment. Approximately 100 weeks.
Description: The SAF (N=333) included all subjects who received any study drug under this protocol.
Groups:
- Aflibercept + Sham PDT: Subjects received 2 milligram (mg) Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period).At Week 12, subjects were assessed for the rescue treatment and randomized to receive Aflibercept injection plus sham photodynamic therapy (only in subjects qualifying for rescue therapy) until Week 52. Between Week 52 and Week 96, the treatment interval could have been extended (typically in increments of 1 or 2 weeks) at the discretion of the investigator when the visual and anatomic outcomes allowed.
- Aflibercept + Active PDT: Subjects received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period). At Week 12, subjects were assessed for the rescue treatment and randomized to receive Aflibercept injection plus active photodynamic therapy (only in subjects qualifying for rescue therapy) until Week 52. Between Week 52 and Week 96, the treatment interval could have been extended (typically in increments of 1 or 2 weeks) at the discretion of the investigator when the visual and anatomic outcomes allowed.
- Aflibercept (Non-randomized): Subjects received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every month for the first 3 months (run-in period), but discontinued study participation before randomization.
Arm/Group | Aflibercept + Sham PDT | Aflibercept + Active PDT | Aflibercept (Non-randomized)
All-Cause Mortality (participants affected / at risk) | 3/157 | 0/161 | 1/15
Serious Adverse Events (participants affected / at risk) | 27/157 | 25/161 | 4/15
Other Adverse Events (participants affected / at risk) | 59/157 | 49/161 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept + Sham PDT (N=157) | Aflibercept + Active PDT (N=161) | Aflibercept (Non-randomized) (N=15)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal pigment epithelial tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Afferent loop syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Senile dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (13) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Transcatheter arterial chemoembolisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept + Sham PDT (N=157) | Aflibercept + Active PDT (N=161) | Aflibercept (Non-randomized) (N=15)
Conjunctival haemorrhage (Eye disorders) | 10 (31) | 5 (8) | 0 (0)
Dry eye (Eye disorders) | 6 (11) | 11 (22) | 0 (0)
Ocular hypertension (Eye disorders) | 3 (4) | 1 (1) | 1 (1)
Visual acuity reduced (Eye disorders) | 7 (7) | 9 (10) | 0 (0)
Vitreous floaters (Eye disorders) | 9 (10) | 1 (1) | 0 (0)
Retinal pigment epithelial tear (Eye disorders) | 4 (4) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 25 (41) | 18 (25) | 0 (0)
Intraocular pressure increased (Investigations) | 6 (18) | 9 (20) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (6) | 13 (13) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less